CLINICAL TRIAL: NCT00179205
Title: Complementary Intradialytic Nutritional Supplementation in Dialysis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding exhausted
Sponsor: Vanderbilt University (Other)
Collaborators: Ross Laboratories (Unknown)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50006
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Nepro nutritional supplement
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nepro nutritional supplement — oral nutritional supplement (1 can) administered during the hemodialysis procedure; every other day, 3 days per week, for 3 months; each can contains a total of 480 calories: 71 calories from protein, 206 calories from carbohydrates and 206 calories from fat.
  Arms: 1
Drug: placebo — oral placebo (1 can) administered during the hemodialysis procedure; every other day, 3 days per week, for 3 months; each can contains a total of 60 calories: 0 calories from protein, 60 calories from carbohydrates, and 0 calories from fat.
  Arms: 2

SUMMARY:
In this study, the investigators hypothesize that long-term administration of adequate intradialytic oral nutritional supplementation will increase visceral protein concentrations and somatic protein stores in malnourished chronic hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. On hemodialysis for more than 6 months
2. Optimally dialyzed with a biocompatible membrane (URR > 70% and/or delivered Kt/V > 1.2)
3. Suboptimal nutritional status identified by:

   * Serum albumin less than or equal to 3.90 g/dl and one of the three following criteria:

     * Protein catabolic rate less than 0.95 g/kg/d calculated by three point urea kinetic modeling on at least 2 occasions over the past 6 months
     * Progressive unintentional weight loss more than 2.5% of the initial or ideal body weight over the past 6 months and/or patients who are less than 90% of standard body weight
     * Biochemical parameters of malnutrition defined by 1 of 2 of the following measurements over the consecutive two months prior to inclusion:

       * Serum transferrin concentration less than 225 mg/dl
       * Serum prealbumin concentration less than 32 mg/dl

Exclusion Criteria:

1. Active auto-immune, inflammatory or infectious disease
2. Documented malignancy within the last 12 months
3. Patients on unusual dietary restrictions
4. Life-expectancy less than 6 months
5. Inability to tolerate nutritional supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
increase in serum albumin | 6 months

SECONDARY OUTCOMES:
increase in lean body mass | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133